CLINICAL TRIAL: NCT01679210
Title: Estudio PARTO: Proyecto pAra Reducir Diabetes Tipo dOs / Project Aiming to Reduce Type twO Diabetes
Brief Title: Study of a Postpartum Diabetes Prevention Program for Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of California, San Diego (Other); Northeastern University (Other); Baystate Medical Center (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lisa Chasan-Taber, Associate Professor of Epidemiology, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH 2R01DK064902-06A1
Record Dates: First submitted 2012-08-07; First posted 2012-09-05 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Experimental): Stage-matched physical activity and diet intervention materials and health education.
  Interventions: Behavioral: Lifestyle Intervention
- Health and Wellness (No Intervention): HW served as the comparison group and received the same number of in-person sessions, telephone calls, and mailings at the same time points as LI. Content was limited to general information available to the public from the ACOG and the American Academy of Pediatrics and did not mention exercise behavior change.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Stage-matched physical activity and diet intervention materials and health education.
  Arms: Lifestyle Intervention

SUMMARY:
The overall goal of this randomized controlled trial is to test the efficacy of a culturally and linguistically modified, individually-tailored lifestyle intervention to reduce risk factors for type 2 diabetes and cardiovascular disease among postpartum Hispanic women with a history of abnormal glucose tolerance during pregnancy.

DETAILED DESCRIPTION:
Specific aims are to evaluate the impact of the intervention on 1) postpartum weight loss, 2) biomarkers associated with insulin resistance (i.e., glucose, insulin, HbA1c, leptin, TNF-α, HOMA, AUCgluc, adiponectin), 3) other cardiovascular risk factors (i.e., blood lipids, blood pressure, CRP, fetuin-A, albumin-to-creatinine ratio), and 4) the adoption and maintenance of postpartum behaviors associated with weight loss and prevention of diabetes risk (i.e., physical activity, diet). Eligible Hispanic women will be recruited after routine GDM screening and randomly assigned to a Lifestyle Intervention (n=150) or a Comparison Health and Wellness (control) intervention (n=150). The intervention will be based on our efficacious exercise and dietary interventions for Hispanics (R01NR011295; WIC Common Pathways). Multimodal contacts (i.e., in-person, telephone counseling, and mailed print-based materials) will be used to deliver the intervention from randomization (29 wks gestation) to 12 months postpartum. Targets of the intervention are to achieve Institute of Medicine Guidelines for postpartum weight loss; American College of Obstetrician and Gynecologist guidelines for physical activity; and American Diabetes Association guidelines for diet. The intervention draws from Social Cognitive Theory and the Transtheoretical Model and addresses the specific social, cultural, economic, and physical environmental challenges faced by underserved Hispanic women. Measures of adherence will include the Pregnancy Physical Activity Questionnaire (PPAQ), accelerometers, and dietary recalls. The project is a Renewal Application of R01 DK064902, a study of lifestyle risk factors for GDM in Hispanic women. The proposed project builds upon the expertise of the investigative team in conducting randomized controlled trials of lifestyle interventions among Hispanic pregnant women (R01 DK074876; S3948 ASPH/CDC) and controlled trials of lifestyle interventions among low-income Hispanics with type 2 diabetes and pre-diabetes (R18 DK0658850; R18DK067549) and can readily be translated into clinical practice in underserved and minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women with one or more glucose values during the diagnostic test meeting or exceeding the thresholds defined according to the American Diabetes Association

Exclusion Criteria:

* history of type 1 or type 2 diabetes, heart disease, or chronic renal disease
* contraindications to postpartum participation in moderate physical activity or a low-fat/high-fiber diet (e.g., Crohn's disease, ulcerative colitis)
* inability to read English or Spanish at a 6th grade level
* <18 or >45 yrs of age
* women carrying multiples

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2013-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Postpartum weight change | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Postpartum weight change will be measured as the difference between weight at 6 or 12 mos postpartum and weight at delivery. Weight will be measured on a digital scale.
Percent of participants meeting postpartum weight goals | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Postpartum weight goals will be defined as weight change to prepregnancy weight if prepregnancy BMI was normal, or a 5% change towards prepregnancy weight if prepregnancy BMI was overweight/obese. Weight will be measured on a digital scale.
Fasting Glucose (FG) | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Fasting Glucose (FG) will be measured enzymatically on the Roche P Modular system using Roche Diagnostics reagents (Indianapolis, IN)(mg/dL).
Fasting Insulin (FI) | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Fasting Insulin (FI) will be measured by an electrochemiluminescence immunoassay on the Roche E Modular system in uU/mL.
Hemoglobin A1c (HbA1c) | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  The Hemoglobin A1c (HbA1c) determination on the Roche P Modular system will be based on turbidimetric immunoinhibition using packed red cells.
Leptin | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Leptin will be measured by an ultra-sensitive ELISA assay, an enzymatically amplified "two-step" sandwich-type immunoassay (R&D Systems, Minneapolis, MN) (pg/mL).
Total Adiponectin | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Total Adiponectin (Multimeric) will be measured using an ELISA method from ALPCO Diagnostics Inc. (Salem, NH).
Lipoprotein Profile | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Lipoprotein Profile: will be simultaneously performed on the Roche P Modular system. Total Cholesterol will be measured enzymatically (mg/dL). Triglycerides will be measured enzymatically with correction for endogenous glycerol (mg/dL). The concentration of High Density Lipoprotein Cholesterol will be determined using a direct enzymatic colorimetric assay (mg/dL). Low Density Lipoprotein Cholesterol will be determined by a homogenous direct method (mg/dL).
High Sensitivity C-Reactive Protein | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  The concentration of High Sensitivity C-Reactive Protein (hsCRP) will be determined using an immunoturbidimetric assay on the Roche P Modular system using reagents and calibrators from DiaSorin (Stillwater, MN) (mg/L).
TNF | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  TNF-receptor II is measured by an ELISA assay from R&D Systems (pg/mL).
Albumin-to-creatinine ratio (ACR) | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Albumin-to-creatinine ratio (ACR): Albumin will be measured by a colorimetric assay, an automated dye-binding method using the Roche P Modular system and Roche Diagnostics reagents (Indianapolis, IN) (g/dL). Creatinine will be measured by an enzymatic method using the Roche P Modular system and Roche Diagnostics reagents (Indianapolis, IN) (mg/dL).
Fetuin-A | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Fetuin-A will be measured by an enzyme immunoassay (EIA) (BioVendor - Candler, NC) (ng/mL).
Physical activity | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Total activity according to intensity will be measured via the Pregnancy Physical Activity Questionnaire (PPAQ) and hip worn accelerometer. (MET-hrs/week).
Dietary Intake | 6 weeks postpartum, 6 months postpartum, 12 months postpartum
  Total calories, along with the other nutrients, will be measured via three 24-hr dietary recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chasan-Taber, ScD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chasan-Taber L, Marcus BH, Rosal MC, Tucker KL, Hartman SJ, Pekow P, Braun B, Moore Simas TA, Solomon CG, Manson JE, Markenson G. Estudio Parto: postpartum diabetes prevention program for hispanic women with abnormal glucose tolerance in pregnancy: a randomised controlled trial - study protocol. BMC Pregnancy Childbirth. 2014 Mar 10;14:100. doi: 10.1186/1471-2393-14-100. PMID 24606590
- [Derived] Wagner KA, St Laurent CW, Pekow P, Marcus B, Rosal MC, Braun B, Manson JE, Whitcomb BW, Sievert LL, Chasan-Taber L. The Impact of a Lifestyle Intervention on Postpartum Cardiometabolic Risk Factors Among Hispanic Women With Abnormal Glucose Tolerance During Pregnancy: Secondary Analysis of a Randomized Trial. J Phys Act Health. 2023 Oct 27;21(1):40-50. doi: 10.1123/jpah.2023-0145. Print 2024 Jan 1. PMID 37890839
- [Derived] Wilkie G, Leung K, Moore Simas TA, Tucker KL, Chasan-Taber L. The Association Between Acculturation and Diet and Physical Activity Among Pregnant Hispanic Women with Abnormal Glucose Tolerance. J Womens Health (Larchmt). 2022 Dec;31(12):1791-1799. doi: 10.1089/jwh.2022.0017. Epub 2022 Aug 30. PMID 36040352
- [Derived] Moore Simas TA, Leung K, Nuss E, Marieni M, Marcus B, Rosal MC, Chasan-Taber L. Factors Associated with Risk of Perinatal Depressive Symptoms Among Puerto Rican Women with Hyperglycemia. Matern Child Health J. 2022 Aug;26(8):1741-1751. doi: 10.1007/s10995-022-03429-y. Epub 2022 Apr 6. PMID 35386031
- [Derived] Hawkins M, Marcus B, Pekow P, Rosal MC, Tucker KL, Spencer RMC, Chasan-Taber L. The Impact of a Randomized Controlled Trial of a Lifestyle Intervention on Sleep Among Latina Postpartum Women. Ann Behav Med. 2021 Aug 23;55(9):892-903. doi: 10.1093/abm/kaaa118. PMID 33580651
- [Derived] Gubrium A, Leckenby D, Harvey MW, Marcus BH, Rosal MC, Chasan-Taber L. Perspectives of health educators and interviewers in a randomized controlled trial of a postpartum diabetes prevention program for Latinas: a qualitative assessment. BMC Health Serv Res. 2019 Jun 6;19(1):357. doi: 10.1186/s12913-019-4207-x. PMID 31170973